CLINICAL TRIAL: NCT05745753
Title: Clinical and Imaging Biomarkers Associated With Plasma ad Cellular Determinants of Cardiovascular Disease at the Time of COVID 19 (CardioCovid)
Brief Title: Clinical and Imaging Biomarkers Associated With Plasma ad Cellular Determinants of Cardiovascular Disease at the Time of COVID 19
Acronym: CARDIOCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pedicino Daniela, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3728
Record Dates: First submitted 2023-02-23; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Cardiovascular Diseases
Keywords: Covid 19; Pneumonia
MeSH Terms: conditions — Cardiovascular Diseases; COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Creation within the data platform of the Cardiology Network of a database of studies containing relevant information on patients with cardiovascular diseases with and without COVID 19; Study the prevalence of cardiovascular risk factors by collecting patient information and analyzing data using conventional statistical analysis and machine learning techniques to develop multivariable models and identify those at greatest risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partecipants with cardiovascular disease (Experimental): The research program will examine imaging and clinical biomarkers associated with plasma and cellular determinants of cardiovascular disease, taking into account the potential effects of COVID-19 infection. This will make it possible to re-evaluate the cardiovascular risk profile of subjects with cardiovascular diseases.
  Interventions: Other: sample blood
- Partecip with cardiovascular disease and affected by COVID-19 (Experimental): In this arm we investigate the immune dysregulation that may play a role in the evolution of cardiovascular disease characteristics of chronic and convalescent COVID-19 participants, in this field we will perform detailed clinical cardiological and immunological phenotyping on enrolled patients.
  Interventions: Other: sample blood

INTERVENTIONS:
Other: sample blood — At the time of enrolment, peripheral blood sampling is expected at the outpatient clinic of the experimental center and the study of the patient's clinical history.
  Other Names: clinical history and peripheral blood sampling

SUMMARY:
Acute and chronic cardiovascular complications of pneumonia are common and result from various mechanisms, including relative ischemia, systemic inflammation, and pathogen-mediated injury. However, there is only limited published data regarding on cardiovascular desease (CV) submissions in the wake of viral outbreaks. Data collected during the COVID-19 pandemic highlighted a number of possible determinants of adverse outcome in these patients, particularly with reference to cardio-respiratory complications.

DETAILED DESCRIPTION:
The risk of death increases substantially after age 60, in men and in overweight patients. Cardiac involvement, characterized by elevation of cardiac Troponin I and brain-like natriuretic peptide, is frequent in COVID-19 patients and is associated with a worse prognosis. Finally, right ventricular (RV) dilatation and dysfunction is the most common echocardiographic abnormality in patients with COVID-19, at least in part due to a substantial incidence of pulmonary thromboembolism (PTE). Cardiac abnormalities in COVID-19 patients include changes in heart rate and cardiac autonomic modulation, as well as systemic activation of inflammatory processes, with endothelial damage and involvement of the CV and respiratory systems.

The research program will examine imaging and clinical biomarkers associated with plasma and cellular determinants of cardiovascular disease, taking into account the potential effects of COVID-19 infection. This will make it possible to re-evaluate the cardiovascular risk profile of subjects with cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Women and men between the ages of 45 and 90;
* Patients diagnosed with cardiovascular disease;
* Patients with diabetes;
* Patients with dyslipidemia;
* Patients with hypertension, myocardial infarction (pre-existing or acute STEMI or NSTEMI event) chronic stable angina, peripheral vascular disease, stroke or TIA

Exclusion Criteria:

* Inflammatory diseases and/or infections (except for the IMA-COVID-19 group);
* Tumors, immunological and/or hematological disorders;
* Ejection fraction less than 40%;
* Treatments with anti-inflammatory drugs, with the exception of low-dose aspirin, and antibiotic therapies up to 1 month before enrolment.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Assess cardiovascular risk | 6 months
  The primary objective is to examine clinical and imaging biomarkers associated with plasma and cellular determinants of cardiovascular disease, taking into account the potential effects of COVID-19 infection, to reevaluate the cardiovascular risk profile of individuals with cardiovascular disease

SECONDARY OUTCOMES:
The prevalence of cardiovascular risk factors in chronic COVID 19 partecipants. | 6 months
  Study the prevalence of cardiovascular risk factors by collecting partecipants information and analyzing data using conventional statistical analysis and machine learning techniques to develop multivariable models and identify those at greatest risk and investigation of immune dysregulation may play a role in the evolution of CV disease characteristics of chronic and convalescent COVID-19 patrtecipants, in this field we will perform detailed clinical cardiological and immunological phenotyping on enrolled patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy